CLINICAL TRIAL: NCT03629470
Title: Effectiveness of Nerve Glide Exercises on Cubital Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-01734
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Cubital Tunnel Syndrome
MeSH Terms: conditions — Cubital Tunnel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): standard conservative treatment
  Interventions: Other: Standard Conservative Treatment
- Group 2 (Experimental): nerve gliding exercises along with the standard conservative treatment.
  Interventions: Other: Standard Conservative Treatment; Other: Nerve Gliding Exercises

INTERVENTIONS:
Other: Standard Conservative Treatment — Range of motion exercises, medication and activity modification.
Other: Nerve Gliding Exercises — Taught by occupational therapist. These exercises involve motions of the wrist, arm and neck. Subjects will be instructed to perform exercises regularly following the occupational therapists' protocol
  Arms: Group 2

SUMMARY:
The objective of this study is to determine if nerve glide exercises in patients with cubital tunnel syndrome can improve pain, paraesthesias and reduce the need for future surgery. Cubital tunnel syndrome is a common form of peripheral neuropathy caused by compression of the ulnar nerve at the elbow. Surgical intervention is typically reserved for those with severe symptoms, but many cases can be treated with non-operative measures. This study will look at the efficacy of nerve glide exercises in the management of cubital tunnel syndrome. 70 subjects with cubital tunnel syndrome will be enrolled and randomized into groups receiving either standard conservative measures or standard measures in addition to nerve glide exercises. Outcomes will be measured 6 months after initiation of treatment with questionnaires on clinical symptoms and function to see if there is a difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with cubital tunnel syndrome on physical exam

Exclusion Criteria:

* Patients with diagnosed or self-reported cognitive dysfunction
* Patients who are unable to understand or follow commands
* Any patient that the investigators feel unsafe or cannot comply with all study related procedures
* Patients who had previous ulnar nerve release at the elbow
* Patients with documented cervical spine pathology
* Patients with clinical signs of other nerve pathology
* Patients with palpable subluxation of the ulnar nerve at the elbow

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Clinical Scoring | 1 Month
  30 item questionnaire used as a clinical scoring system.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Catalano, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No